CLINICAL TRIAL: NCT03517436
Title: A Prospective, Single-arm, Controlled, Multicenter Study to Establish the Safety and Effectiveness of the CENTERA THV System in Intermediate Risk Patients Who Have Symptomatic, Severe, Calcific, Aortic Stenosis Requiring Aortic Valve Replacement
Brief Title: ExCEED: CENTERA THV System in Intermediate Risk Patients Who Have Symptomatic, Severe, Calcific, Aortic Stenosis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-18
Record Dates: First submitted 2018-04-25; First posted 2018-05-07 (Actual); Results first posted 2021-09-30 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Aortic Valve Stenosis
Keywords: THV; Transcatheter Heart Valve; CENTERA; self-expanding
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transcatheter Aortic Valve Replacement (TAVR) (Experimental)
  Interventions: Device: TAVR with CENTERA THV

INTERVENTIONS:
Device: TAVR with CENTERA THV — TAVR with the Edwards CENTERA THV System

SUMMARY:
This study will monitor the safety and valve performance of the Edwards CENTERA Transcatheter Heart Valve (THV) System in patients with symptomatic, severe, calcific aortic stenosis who are at intermediate operative risk for surgical aortic valve replacement (SAVR).

DETAILED DESCRIPTION:
A prospective, single-arm, controlled, multicenter study. Up to 2 roll-ins were allowed per site but not counted towards total enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Severe, calcific AS
2. NYHA functional class ≥ II
3. Judged by the Heart Team to be at intermediate risk for open surgical therapy
4. The subject has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Native aortic annulus size unsuitable for sizes 23, 26 or 29 mm CENTERA THV based on 3D imaging analysis
2. Aortic valve is unicuspid, bicuspid or non-calcified
3. Pre-existing mechanical or bioprosthetic valve in any position
4. Known hypersensitivity to Nitinol (nickel or titanium)
5. Severe aortic regurgitation (> 3+)
6. Severe mitral regurgitation (> 3+) or ≥ moderate stenosis
7. Ventricular dysfunction with left ventricular ejection fraction < 30%
8. Cardiac imaging evidence of intracardiac mass, thrombus or vegetation
9. Evidence of an acute myocardial infarction ≤ 30 days before the valve implant procedure
10. Subjects with planned concomitant ablation for atrial fibrillation
11. Hypertrophic cardiomyopathy with obstruction
12. Coronary anatomy that increases the risk of coronary artery obstruction post-TAVR
13. Complex coronary artery disease
14. Iliofemoral vessel characteristics that would preclude safe placement of the introducer sheath.
15. Significant abdominal or thoracic aortic disease that would preclude safe passage of the delivery system
16. Active bacterial endocarditis within 180 days of the valve implant procedure
17. Stroke or transient ischemic attack within 90 days of the valve implant procedure
18. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis within 30 days of the valve implant procedure
19. Severe lung disease or currently on home oxygen
20. Severe pulmonary hypertension
21. Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation or mechanical heart assistance within 30 days of the valve implant procedure
22. History of cirrhosis or any active liver disease
23. Renal insufficiency and/or renal replacement therapy at the time of screening
24. Leukopenia, anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy or hypercoagulable states
25. Inability to tolerate or condition precluding treatment with antithrombotic therapy during or after the valve implant procedure
26. Absolute contraindications or allergy to iodinated contrast that cannot be adequately treated with pre-medication
27. Significant frailty as determined by the Heart Team
28. Immobility that would prevent completion of study procedures
29. Subject refuses blood products
30. Body mass index > 50 kg/m2
31. Estimated life expectancy < 24 months
32. Positive urine or serum pregnancy test in female subjects of childbearing potential
33. Currently participating in an investigational drug or another device study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2030-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Leon, MD, Principal Investigator — Columbia University Medical Center/ NYPH
Locations (23):
- United States (23):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - UC Health Northern Colorado (Medical Center of the Rockies), Loveland, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - St. Vincent Medical Group, Inc./St. Vincent Heart Center of Indiana, LLC, Indianapolis, Indiana
  - University of Kansas Health System, Kansas City, Kansas
  - Cardiovascular Research Institute of Kansas, Wichita, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Washington University/ Barnes-Jewish Hospital, St Louis, Missouri
  - Atlantic Health System Hospital Corp, Morristown, New Jersey
  - Columbia University Medical Center/ NYPH, New York, New York
  - The Ohio Health Research Institute, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny - Singer Research Institute, Pittsburgh, Pennsylvania
  - Saint Thomas Health, Nashville, Tennessee
  - Baylor Heart and Vascular Hospital, Dallas, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Memorial Hermann, Houston, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas
  - Baylor Scott and White, Central Texas, Temple, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Edwards CENTERA System TAVR: Transcatheter aortic valve replacement (TAVR) with the Edwards CENTERA THV System
Period: Overall Study
Arm/Group | Edwards CENTERA System TAVR
Started | 101
Completed | 93
Not Completed | 8
Not completed — Death | 3
Not completed — Withdrawal by Subject | 4
Not completed — Did not receive study valve. | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Edwards CENTERA System TAVR
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.0 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 91
  More than one race | 1
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: All-cause Death
Description: Number of participants that died
Time Frame: 1 year
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Edwards CENTERA System TAVR
Number analyzed (Participants) | 101
Participants | 3

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Edwards CENTERA System TAVR
All-Cause Mortality (participants affected / at risk) | 3/101
Serious Adverse Events (participants affected / at risk) | 46/101
Other Adverse Events (participants affected / at risk) | 44/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards CENTERA System TAVR (N=101)
Blood loss anaemia (Blood and lymphatic system disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 6 (9)
Atrioventricular block complete (Cardiac disorders) | 11 (11)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 3 (3)
Bundle branch block left (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac failure acute (Cardiac disorders) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardiac perforation (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 2 (2)
Death (General disorders) | 1 (1)
Hernia (General disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (2)
Abdominal wall abscess (Infections and infestations) | 1 (1)
Administration site infection (Infections and infestations) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 3 (4)
Diverticulitis (Infections and infestations) | 1 (1)
Endocarditis bacterial (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Pneumonia bacterial (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (2)
Staphylococcal infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural hypotension (Injury, poisoning and procedural complications) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3)
Metastatic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Intracranial mass (Nervous system disorders) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 3 (3)
Loss of consciousness (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Thalamic infarction (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Device delivery system issue (Product Issues) | 1 (1)
Mental status changes (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Knee arthroplasty (Surgical and medical procedures) | 1 (1)
Femoral artery dissection (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Edwards CENTERA System TAVR (N=101)
Atrial fibrillation (Cardiac disorders) | 10 (11)
Atrioventricular block first degree (Cardiac disorders) | 9 (10)
Bundle branch block left (Cardiac disorders) | 28 (29)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-29): https://cdn.clinicaltrials.gov/large-docs/36/NCT03517436/Prot_SAP_000.pdf